CLINICAL TRIAL: NCT02198625
Title: Influence of Moderate Inspired Oxygen Fraction (FiO2) and Protective Ventilation on Postoperative Pulmonary Complication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fenmei Shi (Other)
Responsible Party: Sponsor-Investigator, Fenmei Shi, resident, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18826410080
Record Dates: First submitted 2014-07-13; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Hepatectomy
Keywords: Moderate FiO2; Protective lung ventilation; Postoperative pulmonary complications; Positive end-expiratory pressure; recruitment maneuvers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FiO2 80%,Nonprotective Lung Ventilation (No Intervention)
- FiO2 30%,Nonprotective Lung Ventilation (Experimental): FiO2 30%,Nonprotective Lung Ventilation
  Interventions: Other: Moderate FiO2 and Protective Lung Ventilation Using
- FiO2 80%,protective Lung Ventilation (Experimental): FiO2 80% and protective Lung Ventilation
  Interventions: Other: Moderate FiO2 and Protective Lung Ventilation Using
- FiO2 30%,protective Lung Ventilation (Experimental): FiO2 30% and protective Lung Ventilation
  Interventions: Other: Moderate FiO2 and Protective Lung Ventilation Using

INTERVENTIONS:
Other: Moderate FiO2 and Protective Lung Ventilation Using
  Arms: FiO2 30%,Nonprotective Lung Ventilation; FiO2 30%,protective Lung Ventilation; FiO2 80%,protective Lung Ventilation

SUMMARY:
The purpose of this study is to determine the influence of moderate FiO2 and the lung protective ventilation on postoperative pulmonary complications following hepatic resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1~2,Planned intrabdominal hepatic resection surgery;
* Expected duration 2 hours to 6 hours;
* Age 40 yr to 70 yr);
* BMI 18-26.9kg/m2
* Risk of postoperative pulmonary complications (Arozullah score ≥2);

Exclusion Criteria:

* Noninvasive ventilation in the last 30 days;
* Recent history of pneumonia, ALI/ARDS (in the last 30 days);
* History of pulmonary resection;
* History of neuromuscular disease;
* Child-Pugh>A grade；
* Patient refusal;

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
a composite of pulmonary and extrapulmonary complications occurring by day 7 after surgery. | during the first seven days after surgery
  The primary outcome was a composite of major pulmonary complications (defined as pneumonia or need for invasive or noninvasive ventilation for acute respiratory failure) and extrapulmonary complications (defined as sepsis, septic shock, or death) within the first 7 days after surgery.

SECONDARY OUTCOMES:
incidence of pulmonary complications | within the 30-day follow-up period
  the incidence of pulmonary complications due to any cause, graded on a scale from 0 (no pulmonary complications) to 4 (the most severe complications);extrapulmonary complications; durations of ICU and hospital stays;
Oxidative stress markers | 2 days
  Oxidative stress markers variation in blood before anesthesia,during and after surgery , and compare with controls.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China